CLINICAL TRIAL: NCT00452465
Title: The ElderCare Project: Primary Healthcare for Community Living Old Elderly
Brief Title: Primary Healthcare for Community Living Old Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Marshal Godwin, Professor, Faculty of Medicine, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 200603MOP-158331-SDA-CJAA
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Care of the Elderly
Keywords: Elderly; Nursing care plan; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A research nurse will meet with participants, complete a detailed nursing assessment and develop of a care plan to help connect participants with resources to allow them to stay in their homes longer.
  Interventions: Behavioral: ElderCare Plan
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: ElderCare Plan — Nursing assessment and development of an appropriate care plan.
  Arms: Intervention

SUMMARY:
Hypothesis: It is hypothesized that older adults who receive the ElderCare intervention will, when compared with a control group of older adults show a significant improvement in quality of life,a significant decrease in symptomatology, significantly higher satisfaction with their care, and less utilization of health care resources.

The Eldercare project involves a detailed assessment by a nurse done in the patients home, followed by the development and delivery of a Eldercare Plan using a Goal Attainment Scaling approach.

Outcomes include quality of life, symptomatology, satisfaction, and health care utilization.

DETAILED DESCRIPTION:
Objectives: The main objective of this study is to improve the care of the old elderly. This will be done by implementing and evaluating a year long program which is intended to optimize quality of life, symptom management and utilization of both health care and community services for the old elderly.

Hypothesis: It is hypothesized that older adults who receive the ElderCare intervention will, when compared with a control group of older adults: a) show a significant improvement in quality of life - as measured by the SF-36, b) show a significant decrease in symptomatology - as measured by the Comorbidity Symptom Scale, c) show significantly higher satisfaction - as measured by the Patient Satisfaction Questionnaire d) have increased utilization of community-based services, e) have fewer emergency room visits, f) have fewer hospitalizations, and g) fewer visits to the family doctor

Research Plan: The ElderCare program is a nurse-based program of home-delivered care that will be linked directly with the primary care practitioner or primary care team of each older adult in the study. The nurse will be part of the primary health care team for a number of different family physicians practices. The nurse will serve as a link or interface between the family physicians practice (or other primary health care professional or team) and the community services. The nurse will i) evaluate the clinical and personal needs of the patient, ii) develop a management plan based on that review (the review includes chart review, patient assessment and contacting community agencies that have been involved with the patients care). , iii)review the plan with the family physician and the patient/family; iv) implement the plan v) provide patient education; and vi) monitor the patient regularly in his/her home over the course of a year. Evaluation will involve comparing a group of old elderly who receive the ElderCare program (intervention) with a control group. Groups will be evaluated using a variety of assessments which will be done at baseline, 6 months and 12 months.

The steps that will be taken in carrying out the research are outlined as follows:

1. Physician Recruitment
2. Patient Recruitment
3. Baseline Data Collection
4. Randomization - Physicians will be cluster randomized to decrease contamination
5. ElderCare Program delivered to intervention group old elderly
6. Usual care for control group old elderly
7. Outcomes measured at 6 and twelve months - outcomes include quality of life, change in symptomatology, patient satisfaction, use of community services, visits to family doctor, hospitalizations, emergency room visits
8. Data Analysis, Interpretation, Reporting and Analysis

ELIGIBILITY:
Inclusion Criteria:

* Patients of a family practice who are 80 years or older, who are independently living and do not have a diagnosis of dementia.

Exclusion Criteria:

* MMSE score 25 or less

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 236 (Actual)
Dates: Start 2007-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Prospective
Symptomology | Prospectiv e
Satisfaction | Prospective
Health care service utilization | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Godwin, MD, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Primary Healthcare Research Unit, Memorial University of Newfoundland, St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Derived] Godwin M, Pike A, McCrate F, Parsons K, Parsons W, Pitcher H, Buehler S, Gadag V, Miller R, Sclater A. The healthy aged: Descriptive analysis by sex of cognitively functioning elderly patients 80 years and older living independently in the community. Can Fam Physician. 2015 Mar;61(3):e142-7. PMID 25932481